## Impact of Aging on Gastrointestinal Permeability During Hyperthermia

Statistical Analysis Plan NCT05816551 October 7, 2024 **Statistical Analysis Plan:** Data will be assessed for model assumptions (i.e., normality, equality of variance) and inspected for influential data points. Non-normally distributed data will be transformed using a log base 10 transformation. Data will be analyzed using linear mixed effect models with main effects of time or trial (within factor) and group (between factor; older vs young) or unpaired t-tests, as appropriate. Statistical significance was set a priori to p < 0.05.